CLINICAL TRIAL: NCT00252070
Title: Fitness and Functional Exercise for People With Arthritis
Brief Title: Fitness and Exercise for People With Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCCDPHP-ASPH3497; ASPH3497
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Arthritis
Keywords: arthritis; exercise; function; pain
MeSH Terms: conditions — Arthritis; Motor Activity; Pain

INTERVENTIONS:
Behavioral: Functional Exercise for People with Arthritis (FEPA)

SUMMARY:
The purpose of this study is to develop and evaluate a progressive, land-based exercise program, that includes muscular and aerobic conditioning, resistance and stabilization exercises and balance training, for persons with arthritis.

DETAILED DESCRIPTION:
There is evidence that people with arthritis who participate in appropriate types of physical activity can improve physical function and pain management. Most existing programs focus on improving flexibility and balance. Less attention has been paid to conditioning and overall functional fitness. To address some of these concerns, this study will develop, evaluate, and implement a non-aquatic physical activity program to increase health-related functional fitness in community-dwelling adults with arthritis. Specific goals are:

1. To develop a systematic and progressive program (FEPA: Functional Exercise for Persons with Arthritis) that integrates muscular and aerobic conditioning, balance and trunk/pelvic stabilization exercises emphasizing joint-protective, multi-plane movement patterns that mimic those used in everyday activities.
2. Implement the FEPA program in an ethnically diverse, low SES community sample of older adults with arthritis.
3. Conduct process, outcomes and impact evaluations to assess the effectiveness of the FEPA program for increasing short- and immediate-term health and functional fitness outcomes.
4. Evaluate the sustainability of the FEPA program through a program logic model process and identify inputs, activities and outputs that contribute to successful program implementation and the building of community capacity to support long-term program maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported doctor-diagnosed arthritis
* No physical limitations precluding exercise participation
* Negative screen for CVD (PAR-Q)
* Age 20+
* English or Spanish speaking

Exclusion Criteria:

* Presence of any condition for which exercise is contraindicated
* Physical inability to complete exercise program

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2005-11; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Six-minute walk
8-foot up-and-go
Arm curl
Back scratch
AIMS-2

SECONDARY OUTCOMES:
Arthritis self-efficacy
Physical activity level
Pain VAS

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Hootman, PhD, Study Chair — Centers for Disease Control and Prevention
Locations (1):
- San Diego State University, San Diego, California, United States